CLINICAL TRIAL: NCT06351410
Title: Assessment of Tear Production, Corneal Staining, and Comfort Level After One Day of Wearing FDA Group I, II, III, IV, and V Contact Lenses Among Pre-Graduate Students at UKM Kuala Lumpur Campus
Brief Title: Assessment of Tear Production, Corneal Staining, and Comfort Level Wearing Different Types of Contact Lenses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JEP 2023-679
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Dry Eye; Dry Eye Syndromes; Contact Lens-induced Corneal Fluorescein Staining
Keywords: Dry Eye; Contact Lens; Corneal Staining; Tears; Comfort
MeSH Terms: conditions — Dry Eye Syndromes; Lacerations

STUDY DESIGN:
Intervention Model Description: 18 participants will be fitted with 2 types of lenses on either eye at one time. There will be a 2-week wash-off period before another 2 set of fittings with another 4 types of lenses.
Masking Description: The 6 types of Contact Lenses used will be labeled as A, B, C, D, E, and F by a co-investigator and will be fitted on the participant's eye randomly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye wearing contact lens (Experimental): The participant will be given two contact lenses (Lens A and B) to be placed on each eye. This phase will be repeated with C &D and lens E & F at different times. Each phase will have a 2 weeks wash-off period
  Interventions: Device: Eye Wearing Contact Lens

INTERVENTIONS:
Device: Eye Wearing Contact Lens — Each participant will be given 2 types of a different group of contact lenses for each eye and need to wear for 8 hours only. Measurements will be done pre and post wearing of lenses

SUMMARY:
This research assesses the tear performance of five distinct types of soft contact lenses commonly found in the market. The study involves contact lens participants, all of whom are students enrolled at UKM. Before the study, participants were instructed to discontinue wearing their usual contact lenses for two weeks. The lenses utilized in this clinical trial all possess current refractive power. Participants are required to wear the lenses for an entire day only. Upon completion of the study, participants will be requested to complete a brief questionnaire.

DETAILED DESCRIPTION:
Before commencing the trial, all participants will undergo an anterior segment examination to ensure the eyes are in a healthy state, free from corneal diseases. Two parameters will be measured during this examination: Tear Break-Up Time (TBUT), which is a non-invasive method used to assess tear break-up, and the Schirmer Test, where a strip is placed on the lower eyelid for five minutes to evaluate tear wetting of the strip.

The level of comfort after wearing contact lenses for 8 hours will be assessed using the Contact Lens Discomfort Index questionnaire.

The sample size is determined using the formula by Daniel (1999). Ten percent of the total sample size represents the number of subjects for this study. Considering a dropout rate of 10%, this study requires 18 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* Age 19-29 years old
* Refractive error is less than -6.00DS with astigmatism is less than -1.00DC
* Have experience wearing Contact Lenses but agree to stop wearing them for 2 weeks before the study starts

Exclusion Criteria:

* smokers (Ward et al. 2010)
* participants with ocular disease or trauma which includes Lasik patients and intra/extraocular surgery.
* pregnant females (Yenerel & Kucumen 2015).
* participants taking medication for systemic diseases (Fraunfelder et al. 2012).

Ages: 19 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05-02 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
To assess the quantity of tears in eyes wearing contact lenses | 5 minutes
  Schirmer Test is done on patients pre and post-wear. Results will be taken after 5 minutes of measurement using Schirmer Strips
To asess the quality of tears in eyes wearing contact lenses | 5 minutes
  NIBUT is done on patients pre and post wear. (10 seconds)
To assess corneal staining in eyes wearing contact lenses | 5 minutes
  Fluorescein in instill at the conjunctiva and staining is observed using cobalt blue light
To assess comfort level of participants using CL Discomfort Index Questionaire | 10 minutes
  8 questions to be answered for each lens

CONTACTS AND LOCATIONS:
Overall Officials: Haliza Abdul Mutalib, PhD, Principal Investigator — National University of Malaysia
Locations (1):
- Optometry Clinic, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Asharlous A, Jafarzadehpur E, Mirzajani A, Khabazkhoob M, Heydarian S, Taghipour A. Tear Deformation Time and optical quality in eyes wearing silicone hydrogel contact lenses. J Curr Ophthalmol. 2016 Jul 25;28(4):226-227. doi: 10.1016/j.joco.2016.07.002. eCollection 2016 Dec. PMID 27830209
- [Background] Brautaset RL, Nilsson M, Leach N, Miller WL, Gire A, Quintero S, Bergmanson JP. Corneal and conjunctival epithelial staining in hydrogel contact lens wearers. Eye Contact Lens. 2008 Nov;34(6):312-6. doi: 10.1097/ICL.0b013e3181891439. PMID 18997539
- [Result] Arroyo-Del Arroyo C, Fernandez I, Lopez-de la Rosa A, Pinto-Fraga J, Gonzalez-Garcia MJ, Lopez-Miguel A. Design of a questionnaire for detecting contact lens discomfort: the Contact Lens Discomfort Index. Clin Exp Optom. 2022 Apr;105(3):268-274. doi: 10.1080/08164622.2021.1896945. Epub 2021 Mar 18. PMID 33735595

DOCUMENTS (1):
  • Study Protocol (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT06351410/Prot_000.pdf